CLINICAL TRIAL: NCT06531681
Title: The Second Affiliated Hospital of Hainan Medical University
Brief Title: Precision Radiotherapy for Tumours Using Magnetic Resonance-guided Linear Accelerator (MR-Linac)
Status: Recruiting | Type: Observational
Sponsor: The Second Affiliated Hospital of Hainan Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-K35-01
Record Dates: First submitted 2024-06-28; First posted 2024-08-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Overall Response Rate; Oncology; Radiation Toxicity; Quality of Life
MeSH Terms: conditions — Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MR-Linac — Radiation therapy with the MR-Linac

SUMMARY:
Aim to observe the application of MR-Linac for precision radiotherapy of tumours, analyse its therapeutic effect, toxic and side effects,Characteristics of dosimetric parameters etc.

DETAILED DESCRIPTION:
Primary endpoint:

· Overall response rate (ORR) : It refers to the proportion of patients whose tumor volume reduction reaches the pre-specified value and can maintain the minimum time requirement, which is a Complete Response (CR) and a partial response (PR). Partial Response) sum of the proportions.

Secondary points:

* Progression-free Survival (PFS) : the time from the start of treatment until objective tumor Progression or all-cause death of the patient.
* Disease Control Rate (DCR) : The percentage of patients whose cancer shrinks or remains stable over time.
* Overall Survival (OS) : the time from the start of treatment to all-cause death.
* Incidence of adverse reactions: toxicity according to Common Toxicity Criteria for Adverse Events (CTCAE).
* Quality of life: The EORTC Quality of Life measure -QLQ-C30-(V3.0) was used, and the higher the score, the higher the quality of life.
* Dosimetric parameters： include gross target volume（GTV）， clinical target volume（CTV），internal target volume(ITV),planning target volume（PTV），γ-passing rate，and limited dose of organs at risk (including average dose, maximum dose, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Patients are undergoing or have undergone imaging or treatment at the MR linac;
* Age 18-75 years, male or female;
* ECOG score 0-2, life expectancy > 6 months;
* Patients provide written informed consent.

Exclusion Criteria:

* Contraindications to MRI, such as claustrophobia and metallic or electronic implants incompatible with MRI;
* The presence of severe comorbidities that, in the opinion of the investigator, · preclude the toleration or completion of radiotherapy;
* Acute inflammatory disease requiring systemic therapy;
* The presence of active infectious disease;
* Pregnant women, nursing mothers, and patients planning to have children during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will receive or have completed imaging or treatment procedures at MR-Linac, Department of Radiotherapy, Second Affiliated Hospital of Hainan Medical University, age 18-75 years, male or female, ECOG score 0-2, life expectancy > 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-08-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 3months， 6months，12months，24months，36months，60months
  The proportion of patients whose tumor volume reduction reached the predetermined value and maintained the minimum time limit requirement was the sum of CR (Complete Response) and PR (Partial Response) proportions.

SECONDARY OUTCOMES:
Progression-Free Survival | 3months， 6months，12months，24months，36months，60months
  The time from the start of treatment until objective tumor Progression or patient all-cause death
Disease Control Rate | 3months， 6months，12months，24months，36months，60months
  The percentage of patients whose cancer shrinks or remains stable over time
Overall survival | 3months， 6months，12months，24months，36months，60months
  Overall survival of participating patients will be obtained from the hospital information systems
Incidence of adverse reactions | 3months， 6months，12months，24months
  Disease-specific toxicity is obtained from the hospital information system. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary
Patient reported Health related quality of life (HRQoL) | 3months，6months，12months，24months
  Patient reported health related quality of life is captured through a questionnaire the Generic European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30. It is a core scale applicable to all cancer patients. It contains a total of 30 items, items 1 to 28 are divided into 4 grades and scored 1 to 4 points, items 29 and 30 are divided into 7 grades and scored 1 to 7 points. The 30 entries are divided into 15 domains, including 5 functional domains (i.e., somatic, role, cognitive, emotional, and social), 3 symptom domains (i.e., fatigue, pain, nausea, and vomiting), 1 quality of life domain, and 6 single entries/domains. A high score on functional or global health status scale represents a high/healthy level of functioning.
Dosimetric parameters：dose of target volume（TV） | During Radiotherapy
  Dose of target volume（TV）includes gross target volume（GTV），clinical target volume（CTV），internal target volume(ITV) and planning target volume（PTV）,Measured by cGy.
Dosimetric parameters：OAR | During Radiotherapy
  Limited dose of organ at risk（OAR） ，includes mean dose（Dmean）, maximum dose（Dmax）and minimum dose（Dmin），Measured by cGy.
  Volume dose limitation，Measured by percent（%），for example， lung V20≤30%.
Dosimetric parameters：γ passing rate | During Radiotherapy
  The gamma passing rate evaluates the coincidence between the calculated and measured dose distributions by utilizing the percent dose difference (DD) and distance to agreement.

CONTACTS AND LOCATIONS:
Overall Officials: yuecan zeng, doctor, Principal Investigator — The Second Affiliated Hospital of Hainan Medical University
Locations (1):
- The Second Affiliated Hospital of Hainan Medical University, Haikou, China